CLINICAL TRIAL: NCT01864057
Title: Pharmacokinetics of Thiamine in Breastfeeding Mothers and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Eastern Mennonite Missions (Unknown); ARUP Laboratories (Other)
Responsible Party: Principal Investigator, Mark Topazian, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MCR 12-004047; NECHR 208
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Beriberi
Keywords: thiamine deficiency
MeSH Terms: conditions — Beriberi; Thiamine Deficiency | interventions — thiamine hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cambodian mothers (Active Comparator): thiamine hydrochloride 100 mg orally daily for 5 days
  Interventions: Drug: thiamine hydrochloride 100 mg
- American mothers (No Intervention): Baseline blood and breast milk sample collection

INTERVENTIONS:
Drug: thiamine hydrochloride 100 mg
  Arms: Cambodian mothers

SUMMARY:
Thiamine deficiency causes beriberi and is common in parts of rural Cambodia, where it appears to be a leading cause of infant death. The change in maternal and infant thiamine level after administration of thiamine to either Cambodian mothers or their infants is unknown. Normal human breast milk thiamine levels in thiamine-replete mothers are poorly characterized. The aim of this study is to determine if thiamine administered to nursing Cambodian mothers normalizes maternal and infant thiamine levels. Levels will also be obtained in nursing Caucasian mothers residing in the United States.

DETAILED DESCRIPTION:
In this pharmacokinetic study, thiamine hydrochloride 100 mg will be administered to nursing Cambodian mothers and thiamine levels will be measured in their blood and breast milk before and after supplementation. Their infant's blood thiamine levels will also be measured. A control arm of American breast feeding mothers taking prenatal vitamins will also be enrolled, to allow comparison of maternal blood and breast milk levels between Cambodian and American mothers. Ethics committee approval was obtained in Cambodia (National Ethics Committee for Health Research #208, 2011) and in the United States (Mayo Clinic Rochester IRB #12-004047)for the Cambodian and American portions of the protocol, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Mother is at least 18 years of age
* Infant is between 1 and 12 months of age
* Cambodian infant is exclusively breast fed
* Cambodian mother has not taken vitamin supplements within the past month
* American mother has been taking prenatal vitamins throughout pregnancy and postpartum while breastfeeding
* Mother and infant do not have an acute illness at the time of enrollment
* Mother and infant are able to comply with study visits

Exclusion Criteria:

* Mother is not able to provide informed consent
* Cambodian infant has received thiamine injections within the past 2 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
blood thiamine concentration | 5 days
  blood thiamine and thiamine diphosphate concentrations after 5 days of maternal oral thiamine supplementation

SECONDARY OUTCOMES:
breast milk thiamine concentration | 5 days
  breast milk thiamine concentration after 5 days of maternal thiamine supplementation

OTHER OUTCOMES:
infant thiamine concentration | 5 days
  infant blood thiamine and thiamine diphosphate concentrations after 5 days of maternal supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Mark Topazian, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Svai Chrum Clinic, Mesang District, Prey Veng, Cambodia

REFERENCES:
- [Background] Coats D, Shelton-Dodge K, Ou K, Khun V, Seab S, Sok K, Prou C, Tortorelli S, Moyer TP, Cooper LE, Begley TP, Enders F, Fischer PR, Topazian M. Thiamine deficiency in Cambodian infants with and without beriberi. J Pediatr. 2012 Nov;161(5):843-7. doi: 10.1016/j.jpeds.2012.05.006. Epub 2012 Jun 14. PMID 22703952
- [Derived] Coats D, Frank EL, Reid JM, Ou K, Chea M, Khin M, Preou C, Enders FT, Fischer PR, Topazian M. Thiamine pharmacokinetics in Cambodian mothers and their breastfed infants. Am J Clin Nutr. 2013 Sep;98(3):839-44. doi: 10.3945/ajcn.113.062737. Epub 2013 Jul 17. PMID 23864540